CLINICAL TRIAL: NCT06986889
Title: COmparison of the HaNd DysFunction in Coronary Diagnosis and INtervention Via Distal vs Conventional Radial AccEss: Randomized Controlled Trial (CONFINE)
Brief Title: Hand Dysfunction in Coronary Diagnosis and Intervention Via Distal Radial Access
Acronym: CONFINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wujin People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20250501
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Coronary Arterial Disease (CAD); Distal Raidal Artery; Hand Functions
Keywords: Coronary arterial disease; Distal radial artery; Conventional radial artery; Hand dysfunction

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-center clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Distal radial artery access group (Experimental): Subjects randomized to experimental group were underwent coronary diagnosis and intervention via distal radial artery access.
  Interventions: Procedure: Distal radial artery access
- Conventional radial artery access group (Active Comparator): Subjects randomized to active comparator group were underwent coronary diagnosis and intervention via conventional radial artery access.
  Interventions: Procedure: Conventional radial artery access

INTERVENTIONS:
Procedure: Conventional radial artery access — Half of the patients enrolled in the study undergoing coronary diagnosis and intervention will be randomized conventional radial access for cardiac catheterization.
  Arms: Conventional radial artery access group
Procedure: Distal radial artery access — Half of the patients enrolled in the study undergoing coronary diagnosis and intervention will be randomized distal radial access for cardiac catheterization.
  Arms: Distal radial artery access group

SUMMARY:
Randomized controlled trial for comparison of the hand dysfunction in coronary diagnosis and intervention via distal vs conventional radial access

DETAILED DESCRIPTION:
Coronary diagnosis and intervention via distal radial access has gradually become an alternative access to the conventional radial access because of its advantages of reducing radial artery occlusion (RAO), shortening compression time, and decreasing patient discomfort. However, as awareness of distal radial access has increased, some patients have been found to have symptoms such as abnormal hand sensation and inflexibility after the procedure.

The primary objective is to assess hand function after coronary diagnosis and intervention via distal vs conventional radial access at 24 hours and 1 month.

Hand sensory and motor dysfunction will be assessed by:

* Consultation and physical examination
* Hand grip test
* Hand pinch test (lateral pinch)
* Monofilament sensory test
* Quick DASH questionnaire
* High-frequent ultrasound The other endpoints include the success rate of puncture, the success rate of single-attempt puncture, time of puncture, procedural duration, duration of hemostasis, vascular complication, etc.

ELIGIBILITY:
Inclusion Criteria

* Indications for coronary diagnosis and intervention
* Distal and conventional radial artery pulsation are palpable
* Patient should be able to comply with the protocol

Exclusion Criteria

* Age < 18 years or ≥ 90 years
* Height ≥ 185 cm
* Acute STEMI
* Haemodynamic instability
* Contraindications to puncture at the puncture site (such as infection, scarring or indwelling needles)
* Enrollment in another study that competes or interferes with this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Hand Numbness | 24 hours after procedure
  Number of participants with the hand numbness is evaluated through clinical consultations at 24 hours after procedure.

SECONDARY OUTCOMES:
Nerve Injury | 24 hours and 1 month after procedure
  Number of participants with the nerve injury is detected using high-frequent ultrasound or electromyography at 24 hours after procedure, and patients with nerve injury at 1 month follow-up will be recorded.
Thumb and Index Finger Pinch Test | 24 hours before and after procedure, 1 month after procedure
  Thumb and forefinger lateral pinch strength (kg)
Hand Grip Test | 24 hours before and after procedure, 1 month after procedure
  Hand grip strength test (kg)
Late-term Hand Numbness | 1 month after procedure
  Number of participants with the hand numbness is evaluated through clinical consultations at 1 month after procedure.
Quick Disabilities of the Arm Shoulder and Hand (DASH) Questionnaire (0-100) | 24 hours before procedure and 1 month after procedure
  Upper extremity dysfunction questionnaire. Scores range from 0 to 100, with higher scores indicating greater dysfunction.
Visual Analogue Scale (VAS) Scale (0-10) | 24 hours after procedure
  Pain assessment. Scores range from 0 to 10, with higher scores indicating greater pain intensity.
Hand Paresthesia | 24 hours and 1 month after procedure
  Number of participants with the hand paresthesia is assessed using monofilament test and/or two-point discrimination test at 24 hours after procedure, and patients with hand paresthesia at 1 month follow-up will be recorded.
Hand Clumsiness | 24 hours and 1 month after procedure
  Number of participants with the hand clumsiness at 24 hours after procedure, and patients with hand clumsiness at 1 month follow-up will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Cai, MD, Study Chair — Cardiovascular department, Changzhou Wujin People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Leeuwen MA, van Mieghem NM, Lenzen MJ, Selles RW, Hoefkens MF, Zijlstra F, van Royen N. The effect of transradial coronary catheterization on upper limb function. JACC Cardiovasc Interv. 2015 Apr 20;8(4):515-23. doi: 10.1016/j.jcin.2014.10.025. Epub 2015 Mar 26. PMID 25819177
- [Background] Sgueglia GA, Hassan A, Harb S, Ford TJ, Koliastasis L, Milkas A, Zappi DM, Navarro Lecaro A, Ionescu E, Rankin S, Said CF, Kuiper B, Kiemeneij F. International Hand Function Study Following Distal Radial Access: The RATATOUILLE Study. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1205-1215. doi: 10.1016/j.jcin.2022.04.023. Epub 2022 May 17. PMID 35595672
- [Background] Tehrani BN, Sherwood MW, Damluji AA, Epps KC, Bakhshi H, Cilia L, Dassanayake I, Eltebaney M, Gattani R, Howard E, Kepplinger D, Ofosu-Somuah A, Batchelor WB. A Randomized Comparison of Radial Artery Intimal Hyperplasia Following Distal Versus Proximal Transradial Access for Coronary Angiography: PRESERVE RADIAL. J Am Heart Assoc. 2024 Feb 20;13(4):e031504. doi: 10.1161/JAHA.123.031504. Epub 2024 Feb 14. PMID 38353242
- [Background] Daralammouri Y, Nazzal Z, Mosleh YS, Abdulhaq HK, Khayyat ZY, Hamshary YE, Azamtta M, Ghanim A, Awwad F, Majadla S, Maree M, Hamaida J, Ismail Y. Distal Radial Artery Access in comparison to Forearm Radial Artery Access for Cardiac Catheterization: A Randomized Controlled Trial (DARFORA Trial). J Interv Cardiol. 2022 Jul 15;2022:7698583. doi: 10.1155/2022/7698583. eCollection 2022. PMID 35911661
- [Background] Chen T, Li L, Li F, Lu W, Shi G, Li W, Yang A, Huang H, Xiao J, Zhang Q, Gu J, Xue S, Zhang L, Li L, Xu L, Ji R, Wang H, Cai G. Comparison of long-term radial artery occlusion via distal vs. conventional transradial access (CONDITION): a randomized controlled trial. BMC Med. 2024 Feb 8;22(1):62. doi: 10.1186/s12916-024-03281-7. PMID 38331793
- [Background] Babunashvili AM, Pancholy S, Zulkarnaev AB, Kaledin AL, Kochanov IN, Korotkih AV, Kartashov DS, Babunashvili MA. Traditional Versus Distal Radial Access for Coronary Diagnostic and Revascularization Procedures: Final Results of the TENDERA Multicenter, Randomized Controlled Study. Catheter Cardiovasc Interv. 2024 Dec;104(7):1396-1405. doi: 10.1002/ccd.31271. Epub 2024 Oct 30. PMID 39474765
- [Background] Aminian A, Sgueglia GA, Wiemer M, Kefer J, Gasparini GL, Ruzsa Z, van Leeuwen MAH, Ungureanu C, Leibundgut G, Vandeloo B, Kedev S, Bernat I, Ratib K, Iglesias JF, Al Hage E, Posteraro GA, Pascut D, Maes F, Regazzoli D, Kakonyi K, Meijers TA, Colletti G, Krivoshei L, Lochy S, Zafirovska B, Horak D, Nolan J, Degrauwe S, Tobita K, Saito S. Distal Versus Conventional Radial Access for Coronary Angiography and Intervention: The DISCO RADIAL Trial. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1191-1201. doi: 10.1016/j.jcin.2022.04.032. Epub 2022 May 17. PMID 35595673
- [Background] Al-Azizi K, Moubarak G, Dib C, Sayfo S, Szerlip M, Thomas S, Hale S, Zyl JV, Settele RM, Gonzalez OR, Ventura SJ, DiMaio JM, Mack MJ, Potluri S. Distal Versus Proximal Radial Artery Access for Cardiac Catheterization: 1-Year Outcomes. Am J Cardiol. 2024 Jun 1;220:102-110. doi: 10.1016/j.amjcard.2024.02.036. Epub 2024 Mar 2. PMID 38432334
- [Background] Kozinski L, Orzalkiewicz Z, Dabrowska-Kugacka A. Feasibility and Safety of the Routine Distal Transradial Approach in the Anatomical Snuffbox for Coronary Procedures: The ANTARES Randomized Trial. J Clin Med. 2023 Dec 11;12(24):7608. doi: 10.3390/jcm12247608. PMID 38137677
- [Background] Gupta M, Kumar V, Rahman MW, Srivastava S, Pandey U, Sinha SK. Comparison Between Distal Trans-radial Access and Conventional Trans-radial Access for Coronary Angiography. Cureus. 2023 Sep 12;15(9):e45081. doi: 10.7759/cureus.45081. eCollection 2023 Sep. PMID 37842393